CLINICAL TRIAL: NCT05542446
Title: Pharmacokinetics of Colistin in Critically Ill Patients With Extracorporeal Membrane Oxygenation
Acronym: COL-ECMO2022
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: After agreement between sponsor and investigator, insufficient patients recruitment
Sponsor: St. Anne's University Hospital Brno, Czech Republic (Other)
Collaborators: Palacky University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: COL-ECMO2022; 2022-000291-19 (EudraCT Number)
Record Dates: First submitted 2022-08-18; First posted 2022-09-15 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Colistin
Keywords: colistin; critically ill; pharmacokinetics; extracorporeal membrane oxygenation; investigator-initiated study
MeSH Terms: conditions — Critical Illness | interventions — Colistin; colistinmethanesulfonic acid

STUDY DESIGN:
Intervention Model Description: The primary objective of the clinical trial is to determine the plasma concentrations of colistin and CMS during the one or more monitored dosing interval(s) in critically ill patients with and without ECMO under the real clinical practice conditions; based on these data to calculate and compare the pharmacokinetic parameters (Cmax, Tmax, Ctrough, AUC, Vd, clearance) of CMS and colistin in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Critically ill patients with ECMO (Experimental): The subjects connected to ECMO will be treated with colistin ain approved dosing - a loading dose of 9 MIU intravenously over 30 minutes followed after 12 hours by a maintenance dose of 4,5 MIU intravenously over 30 minutes every 12 hours. Only in patients requiring continuous renal replacement methods will the interval of the maintenance doses be 8 hours.
  Interventions: Drug: Colistin
- Critically ill patients without ECMO (Active Comparator): The subjects not connected to ECMO will be treated with colistin ain approved dosing - a loading dose of 9 MIU intravenously over 30 minutes followed after 12 hours by a maintenance dose of 4,5 MIU intravenously over 30 minutes every 12 hours. Only in patients requiring continuous renal replacement methods will the interval of the maintenance doses be 8 hours.
  Interventions: Drug: Colistin

INTERVENTIONS:
Drug: Colistin — Visit 1 - screening - Patient selection phase. Patients meeting the eligibility criteria will be screened if not meeting any of the exclusion criteria. A pregnancy test from a urine test will be performed on women of childbearing potential. The patient will be offered participation in the clinical trial and interviewed by the investigator.
  Visit 2 (Visit 8, Visit 14 - optional, only if colistin is still indicated) - CMS administration The patient will be hospitalized at FNUSA. CMS will be given intravenously via the central vein catheter (a loading dose of 9 MIU intravenously over 30 minutes followed after 12 hours by a maintenance dose of 4,5 MIU intravenously over 30 minutes every 12 hours; only in patients requiring continuous renal replacement methods will the interval of the maintenance doses be 8 hours).
  Visit 3 - Visit 7 (Visit 9-Visit 13, Visit 15-Visit 19 - optional, only if colistin is still indicated) - Pharmacokinetics blood samples collection.
  Other Names: colistin methanesulfonate; colistimethate

SUMMARY:
Colistin is a lipopeptide antibiotic administered as an inactive prodrug - colistin methanesulfonate (CMS). Colistin is a drug with a narrow therapeutic window; the limiting factors are mainly nephrotoxicity and neurotoxicity dependent on plasma concentrations. The number of patients with these types of infections, as well as the number of patients requiring extracorporeal membrane oxygenation (ECMO) support for severe respiratory failure, increased significantly in association with COVID-19-induced infections. ECMO can generally affect the pharmacokinetics of drugs by creating a new compartment.

DETAILED DESCRIPTION:
The COL-ECMO2022 study is a prospective, non-randomized, open-label single-center, phase IV clinical trial that is designed to assess the influence of ECMO on the pharmacokinetics of colistin and CMS. The study is planned to include up to 30 patients with indication of colistin who will be assigned to one of two arms in a 1:1 ratio depending on the presence/absence of ECMO. All study participants will receive colistin standard, approved dose schedule intravenously. The plasma concentrations of colistin and CMS took at defined intervals will be assessed by high-performance liquid chromatography-mass spectrometry. Patients will participate in the clinical trial for a maximum of three monitored dosing intervals.

Discussion: This study is expected to provide essential evidence-based data on the impact of ECMO on colistin pharmacokinetics in critically ill patients as well as to shed some light on how to optimize the colistin dosing for critically ill patients on ECMO by designing the population model.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Men and women (with a negative pregnancy test prior to study enrolment in women of childbearing potential)
* Hospitalized at the Department of Anaesthesiology and Resuscitation, St. Anne´s University Hospital Brno
* Indication for parenteral colistin (or CMS) as part of standard medical care, i.e., in patients with severe bacterial infection
* Informed consent given. In unconscious patients, the study investigator will decide whether to include the patient in the study; this decision is made whenever possible in a medical council consisting of at least one independent physician informed about the study details and one study investigator. An interim informed consent will be given after considering all individual risks. In this case, the Ethics Committee of St. Anne's Hospital in Brno will be informed of the patient's inclusion. The investigator will ask study participants in whom good quality consciousness is restored to give subsequent informed consent without unreasonable delay.

Additional inclusion criterion:

For some patients (15 individuals are expected), in addition to all the criteria listed in the Eligibility Criteria section, the following inclusion criterion is provided:

* ECMO support is needed as part of standard therapy for severe respiratory failure.

Exclusion Criteria:

* Pregnancy,
* Breast-feeding,
* Refusal to give the informed consent (primarily or after regaining consciousness).

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Verification of the ECMO-induced changes of colistin or CMS area under the plasma concentration versus time curve (AUC) in critically ill patients. | 24 hours
  The primary objective of the clinical trial is to determine the area under the plasma concentration versus time curve of colistin and CMS in critically ill patients with and without ECMO during the dosing interval, calculate and compare the area under the plasma concentration versus time curve of CMS and colistin in each group.

SECONDARY OUTCOMES:
Model of population pharmacokinetics of colistin in critically ill patients - Cmax | 2 hours after colistin administration. The model will be designed through study completion, an average of 1 year
  To propose a model of population pharmacokinetics of colistin in critically ill patients. The pharmacokinetic model will be designed as a composite of several pharmacokinetics parameters that will be obtained during the individual measurements. The first one is maximum plasma concentrations [Cmax] that will be obtain 2 hours after colistin administration.
Model of population pharmacokinetics of colistin in critically ill patients - Tmaxc | 2 hours after colistin administration. The model will be designed through study completion, an average of 1 year
  To propose a model of population pharmacokinetics of colistin in critically ill patients. The pharmacokinetic model will be designed as a composite of several pharmacokinetics parameters that will be obtained during the individual measurements. The second one is time to maximum plasma concentration (Tmaxc) that will be calculated within 2 hours after colistin administration.
Model of population pharmacokinetics of colistin in critically ill patients - Tminc | 12 hours after colistin administration. The model will be designed through study completion, an average of 1 year
  To propose a model of population pharmacokinetics of colistin in critically ill patients. The pharmacokinetic model will be designed as a composite of several pharmacokinetics parameters that will be obtained during the individual measurements. The third one is time to minimum plasma concentration (Tminc) that will be calculated within 12 hours after colistin administration.
Model of population pharmacokinetics of colistin in critically ill patients - Cmin | 12 hours after colistin administration. The model will be designed through study completion, an average of 1 year
  To propose a model of population pharmacokinetics of colistin in critically ill patients. The pharmacokinetic model will be designed as a composite of several pharmacokinetics parameters that will be obtained during the individual measurements. The fourth one is minimum plasma concentration (Cmin) that will be calculated within 12 hours after colistin administration.
Model of population pharmacokinetics of colistin in critically ill patients - AUC | 24 hours after colistin administration. The model will be designed through study completion, an average of 1 year
  To propose a model of population pharmacokinetics of colistin in critically ill patients. The pharmacokinetic model will be designed as a composite of several pharmacokinetics parameters that will be obtained during the individual measurements. The fifth one is Area Under the Curve (AUC) that will be calculated within 24 hours after colistin administration.

CONTACTS AND LOCATIONS:
Overall Officials: Lucie Tesárková, Scs., Study Chair — St. Anne´s University Hospital Brno
Locations (1):
- St. Anne's University Hospital Brno, Brno, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suk P, Rychlickova J, Souckova L, Kubickova V, Urbanek K. Changes of colistin pharmacokinetics in critically ill patients due to the extracorporeal membrane oxygenation: protocol for the COL-ECMO2022 trial - a prospective, non-randomised, open-label phase IV pharmacokinetic clinical trial. BMJ Open. 2023 Jul 30;13(7):e071649. doi: 10.1136/bmjopen-2023-071649. PMID 37518089